CLINICAL TRIAL: NCT00348439
Title: A Multicenter, Randomized, Double Masked, Placebo Controlled, Sequential Dose Response Study of Intravitreally Administered Plasmin for the Creation of a Posterior Vitreous Detachment (PVD)
Brief Title: Study to Evaluate Plasmin for the Creation of a Posterior Vitreous Detachment
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Lack of Efficacy
Sponsor: Bausch & Lomb Incorporated (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 437
Record Dates: First submitted 2006-06-30; First posted 2006-07-04 (Estimated); Last update posted 2019-06-21 (Actual); Status verified 2019-06

CONDITIONS: Vitreoretinal Traction Syndrome
MeSH Terms: interventions — Fibrinolysin

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Plasmin Injection (Experimental): human-derived plasmin
  Interventions: Drug: Plasmin
- Vehicle (Placebo Comparator): Plasmin formulation, without active ingredient.
  Interventions: Drug: Vehicle

INTERVENTIONS:
Drug: Plasmin — 27 mg of human-derived plasmin to be reconstituted with 0.9% Sterile Sodium Chloride for a single intravitreal injection.
  Arms: Plasmin Injection
Drug: Vehicle — Plasmin formulation, without active ingredient to be reconstituted in 0.9% Sterile Sodium Chloride and administered in a single intravitreal injection.
  Arms: Vehicle

SUMMARY:
Plasmin is expected to create a posterior vitreous detachment. The pharmacological creation of a posterior vitreous detachment may be beneficial in a variety of conditions.

ELIGIBILITY:
Inclusion Criteria:

* Patients who would benefit from a posterior vitreous detachment, as determined by the evaluating ophthalmologist.

Exclusion Criteria:

* Presence of a posterior vitreous detachment in the study eye
* History of vitrectomy in the study eye
* Proliferative diabetic retinopathy in the study eye
* Presence of media opacity that precludes quality examination of the vitreous and fundus.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 29 (Actual)
Dates: Start 2006-04; Primary Completion 2007-08 (Actual); Study Completion 2007-08 (Actual)

PRIMARY OUTCOMES:
Presence of a Grade A Posterior Vitreous Detachment (PVD) | 14 Days
  PVD at the disc and macula post plamin injection

CONTACTS AND LOCATIONS:
Locations (1):
- Emory University, Atlanta, Georgia, United States